CLINICAL TRIAL: NCT03039946
Title: Automated Closed-Loop Versus Restrictive Fluid Therapy in Abdominal Surgery: a Pilot Randomized Controlled Trial
Brief Title: Automated Closed-Loop Versus Restrictive Fluid Therapy in Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P2016/526
Record Dates: First submitted 2017-01-31; First posted 2017-02-01 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-01

CONDITIONS: Abdominal Laparoscopic and/or Robotic Surgery
Keywords: Fluid therapy; Hemodynamic flow monitoring; Closed-loop system; Goal-directed fluid therapy; Anesthesiology

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Closed-loop GDFT (Experimental): This group consists of patients undergoing laparoscopic and/or robotic abdominal surgery where fluid maintenance with Plasmalyte is carried out using a closed-loop system guided by the Clearsight non-invasive hemodynamic flow monitor.
  Interventions: Device: Closed-Loop GDFT
- Restrictive fluid therapy (Active Comparator): This group consists of patients undergoing laparoscopic and/or robotic abdominal surgery where fluid management is based on a restrictive (4ml/kg/h) Plasmalyte infusion.
  Interventions: Other: Restrictive Fluid Therapy

INTERVENTIONS:
Device: Closed-Loop GDFT — Patients receive fluids in the form of 100ml boluses of crystalloid (Plasmalyte) over 6 minutes via an automated closed-loop goal-directed fluid therapy (GDFT) system guided by non-invasive flow monitoring (Clearsight system). Additional boluses of colloid or crystalloid can be administered under the attending anesthesiologist's discretion (e.g. to compensate blood loss) .
  Arms: Closed-loop GDFT
Other: Restrictive Fluid Therapy — Patients receive fluids (Plasmalyte) via a restrictive approach with a baseline of of 4ml/kg/h. Additional boluses of colloid or crystalloid can be administered under the attending anesthesiologist's discretion (e.g. to compensate blood loss) .
  Arms: Restrictive fluid therapy

SUMMARY:
The aim of this study is to compare hemodynamic variables and outcome in patients undergoing laparoscopic and/or robotic elective abdominal surgery. Patients will receive either an automated closed-loop goal-directed fluid therapy (GDFT) guided by non-invasive flow monitoring or a restrictive fluid therapy of 4ml/kg/h.

DETAILED DESCRIPTION:
Perioperative fluid management is a topic of much debate that has intensified over recent years. Studies have shown improved postoperative outcomes with restricted fluid administration in the perioperative period for moderate risk abdominal surgery. They concluded that in patients undergoing elective abdominal surgery, intraoperative restrictive fluid management was associated with a reduction in postoperative morbidity and shortened hospital stay. Current standard practice is a crystalloid based fluid therapy guided by static hemodynamic parameters such as heart rate, blood pressure, and diuresis. However, several studies have criticized this cookbook approach and recommend tailoring management to specific physiologic dynamic endpoints such as stroke volume variation and cardiac output using a flow monitoring device. Our team has demonstrated that the use of a closed-loop system is feasible and allows precise titration of fluid administration in abdominal and vascular surgery using either a minimally or a non-invasive monitoring system.

Goal:

This study compares hemodynamic variables and outcome in patients who will receive either automated closed-loop fluid therapy guided by non-invasive flow monitoring or restrictive fluid therapy of 4ml/kg/h. Both groups consist of the same population undergoing laparoscopic and/or robotic surgery.

Hypothesis:

A closed-loop assisted intraoperative GDFT when compared to restrictive fluid therapy will provide better hemodynamic variables.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic and/or robotic elective abdominal surgery( colorectal, gynecological, urological)

Exclusion Criteria:

* Intraoperative invasive monitoring (arterial line)
* Open colorectal surgery (laparotomy)
* Emergency surgery
* Expected intraoperative blood loss greater than 1000ml
* Arrhythmia (e.g. atrial fibrillation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Preload independent state | 6 hours
  The percentage intraoperative time spent with stroke volume variation < 13% and/or cardiac index > 2.4 L/min/m2

SECONDARY OUTCOMES:
Additional fluids administered intraoperatively | 6 hours
Number of closed-loop override by the attending anesthesiologist | 6 hours
Hospital length of stay | up to 90 days post surgery
Postoperative complications | up to 90 days after hospitalization
  Major complications include cardiac (acute coronary syndrome/ arrhythmia), pulmonary (embolism/edema), gastrointestinal (bowel and surgical anastomotic leak/internal or external fistulas/peritoneal effusions), renal (renal failure requiring dialysis), infectious (peritonitis/ sepsis), coagulation (bleeding), wound dehiscence, stroke, reoperation, readmission, and death.
  Minor complications include unplanned ICU admission, pneumonia/pleural effusion, deep venous thrombosis, paralytic ileus, renal insufficiency, infection (superficial wound infection/fever/urinary infection) and confusion/delirium.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasme University Hospital, Brussels, Belgium

REFERENCES:
- [Background] Donati A, Loggi S, Preiser JC, Orsetti G, Munch C, Gabbanelli V, Pelaia P, Pietropaoli P. Goal-directed intraoperative therapy reduces morbidity and length of hospital stay in high-risk surgical patients. Chest. 2007 Dec;132(6):1817-24. doi: 10.1378/chest.07-0621. Epub 2007 Oct 9. PMID 17925428
- [Background] Giglio MT, Marucci M, Testini M, Brienza N. Goal-directed haemodynamic therapy and gastrointestinal complications in major surgery: a meta-analysis of randomized controlled trials. Br J Anaesth. 2009 Nov;103(5):637-46. doi: 10.1093/bja/aep279. PMID 19837807
- [Background] Rinehart J, Lilot M, Lee C, Joosten A, Huynh T, Canales C, Imagawa D, Demirjian A, Cannesson M. Closed-loop assisted versus manual goal-directed fluid therapy during high-risk abdominal surgery: a case-control study with propensity matching. Crit Care. 2015 Mar 19;19(1):94. doi: 10.1186/s13054-015-0827-7. PMID 25888403
- [Derived] Joosten A, Raj Lawrence S, Colesnicenco A, Coeckelenbergh S, Vincent JL, Van der Linden P, Cannesson M, Rinehart J. Personalized Versus Protocolized Fluid Management Using Noninvasive Hemodynamic Monitoring (Clearsight System) in Patients Undergoing Moderate-Risk Abdominal Surgery. Anesth Analg. 2019 Jul;129(1):e8-e12. doi: 10.1213/ANE.0000000000003553. PMID 29878939